CLINICAL TRIAL: NCT05673265
Title: Pediatric and Adult Registry for Patients With ARThrogryposis
Acronym: PARART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC21.055
Record Dates: First submitted 2022-09-20; First posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-06

CONDITIONS: Arthrogryposis Multiplex Congenita (AMC)
MeSH Terms: conditions — Arthrogryposis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is Epidemiological Evaluation of a single-centre national cohort of patients with Arthrogryposis multiplex congenita (AMC)

DETAILED DESCRIPTION:
Arthrogryposis multiplex congenita (AMC) is a group of rare diseases characterized by joint limitation at least two distinct articular levels at birth which represents about 100 to 200 births with AMC in France per year.

The Reference Center (CR) at Grenoble Alpes University Hospital set up multidisciplinary consultations for pediatric and adult patients with AMC such as (MPR, orthopedics, genetics for children and adults, and pulmonologist, rheumatologist for adults , also including individual or group therapeutic education sessions) .

For develop the diagnostic and follow-up approach, the Reference center initiated the drafting of a diagnostic and care protocol (PNDS), on the one hand based on the data of the literature and on the other hand on expert opinions.

The project is based on four elements :

1. This project is pediatric and adult registry. It should be possible to obtain more comprehensive prognostic data, particularly in relation to complications and possible comorbidities related to older ages.
2. The Recruitment of the patient is done immediately in France who's followed at the reference center in Grenoble Alpes University Hospital.

3-There are several ways for patient addressing. Indeed these are also addressed by the professionals or patients contact the center directly

4-The Patient's assessments are multidisciplinary from the outset, this should lead to get comprehensive functional and diagnostic data.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with arthrogryposis multiplex congenita prenatally or postnatally seen at least once at the reference center from January 2008 to July 2023.
2. pediatric and adult individuals.
3. Addressed to the reference centre of the University Hospital Grenoble Alpes.
4. living in France.

Exclusion Criteria:

1. Individuals who did not consent to use their data (or the data of their children).
2. Individuals with less than two affected joint levels.
3. Individuals under guardianship or deprived of liberty.
4. Inability to collect comprehensive medical information (individuals recently arrived in France)

Max Age: 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult individuals are addressed to the reference centre of the University Hospital Grenoble Alpes for arthrogryposis multiplex congenita (AMC). The assessment is based on multidisciplinary consultations (physical medicine and rehabilitation, orthopedics, genetics for children and adults, and pulmonologist, rheumatologist for adults). The aim of the study is to obtain more comprehensive prognostic data, particularly in relation to complications and possible comorbidities related to older ages.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of etiologies | 2 years
  The etiologies will be drawn up either by the confirmation of a genetic cause by a high-throughput sequencing analysis (NGS), a chromosomal analysis on a DNA chip (ACPA) and / or a leukocyte karyotype, or on anamnestic, clinical and paraclinical data for entities currently without genetic cause retained

SECONDARY OUTCOMES:
Data from complementary examinations (molecular analyses) | 2 years
  Data from complementary examinations (molecular analyses); patients admitted since 2008 to ensure the quality and completeness of the data collected on the historical cohort)
Data from complementary examinations ( medical imaging including muscular MRI) | 2 years
  Data from complementary examinations ( medical imaging including muscular MRI); patients admitted since 2008 to ensure the quality and completeness of the data collected on the historical cohort)
Data from complementary examinations(biochemical analyses) | 2 years
  Data from complementary examinations ( biochemical analyses); patients admitted since 2008 to ensure the quality and completeness of the data collected on the historical cohort)
Data from complementary examinations (pathology) | 2 years
  Data from complementary examinations (pathology); patients admitted since 2008 to ensure the quality and completeness of the data collected on the historical cohort)
Results of phenotypic and functional assessment | 2 years
  Physical examination
Results of phenotypic and functional assessment | 2 years
  Antenatal data
Results of phenotypic and functional assessment | 2 years
  Medical Research Council(MRC) score for muscle strength
Results of phenotypic and functional assessment | 2 years
  Goniometry for joint involvement
Results of phenotypic and functional assessment | 2 years
  Measurement of functional independence(FIM)
Number and types of surgical procedures | 2 years
  Number and types of surgical procedures

CONTACTS AND LOCATIONS:
Overall Officials: Klaus DIETERICH, MD, PhD, Principal Investigator — Univ. Grenoble Alpes Inserm U1209 IAB CHU Grenoble Alpes
Locations (1):
- CHU Grenoble Alpes, La Tronche, France

IPD SHARING:
Plan to Share IPD: No